CLINICAL TRIAL: NCT03570983
Title: A Trial Comparing Single Agent Melphalan to Carmustine, Etoposide, Cytarabine and Melphalan (BEAM) as a Preparative Regimen for Patients With Multiple Myeloma Undergoing High Dose Therapy Followed by Autologous Stem Cell Reinfusion
Brief Title: A Trial Comparing Single Agent Melphalan to Carmustine, Etoposide, Cytarabine, and Melphalan (BEAM) as a Preparative Regimen for Patients With Multiple Myeloma Undergoing High Dose Therapy Followed by Autologous Stem Cell Reinfusion
Acronym: BEAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY2017000117
Record Dates: First submitted 2018-06-08; First posted 2018-06-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Allopurinol; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BEAM Regimen- Experimental Arm (Experimental): Allopurinol Dosage: Allopurinol 200 mg/m2/day starts on the day prior to BCNU, day -8 and stops on day -1.
  BCNU (Carmustine) Dosage: Carmustine 300 mg/m2 IV x 1 will be infused over 3 hours on autografting day -7. Carmustine should not be infused with solutions or tubing containing or previously containing bicarbonate solution.
  Etoposide (VP-16, Vepesid) Dosage: Etoposide 100 mg/m2 IV BID will be administered in 500-1000 cc normal saline over 2 hours on autografting days -6, -5, -4, and -3 for a total dose of 800 mg/m2. Etoposide may not be infused with sodium bicarbonate solutions.
  Cytarabine (Ara-C) Dosage: Cytarabine 100 mg/m2 IV BID will be infused over 3 hours on autografting days -6, -5, -4 and -3.
  Interventions: Drug: Allopurinol; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine
- Melphalan Regimen- Control Arm (Active Comparator): Melphalan Dosage: Melphalan will be administered at a dose of 200 mg/m2 IV x 1 infused over 30 minutes on autografting day -2.
  Allopurinol Dosage: Allopurinol 200 mg/m2/day starts on the day prior to melphalan (day -3) and stops on day -1.
  Interventions: Drug: Allopurinol; Drug: Melphalan

INTERVENTIONS:
Drug: Allopurinol — Dosage: Allopurinol 200 mg/m2/day starts on the day prior to BCNU, day -8 and stops on day -1.
Drug: Carmustine — Dosage: Carmustine 300 mg/m2 IV x 1 will be infused over 3 hours on autografting day -7. Carmustine should not be infused with solutions or tubing containing or previously containing bicarbonate solution.
  Arms: BEAM Regimen- Experimental Arm
Drug: Etoposide — Dosage: Etoposide 100 mg/m2 IV BID will be administered in 500-1000 cc normal saline over 2 hours on autografting days -6, -5, -4, and -3 for a total dose of 800 mg/m2. Etoposide may not be infused with sodium bicarbonate solutions.
  Arms: BEAM Regimen- Experimental Arm
Drug: Cytarabine — Dosage: Cytarabine 100 mg/m2 IV BID will be infused over 3 hours on autografting days -6, -5, -4 and -3. Availability and administration: Cytarabine is available in a reconstituted form in solutions containing 20, 50 and 100 mg of cytarabine per mL.
  Arms: BEAM Regimen- Experimental Arm
Drug: Melphalan — Melphalan will be administered at a dose of 200 mg/m2 IV x 1 infused over 30 minutes on autografting day -2.
  Arms: Melphalan Regimen- Control Arm

SUMMARY:
The work proposed herein aims to provide the first prospective, randomized comparative efficacy data between Melphalan and BEAM treatment regimen in the Multiple Myeloma (MM) patient population. The risk of such a study is deemed reasonable and ethical since: a) previous works have closely examined the safety and toxicity of the BEAM regimen and the doses to be delivered in this protocol are well below the toxicity levels; b) phase III trials of BEAM have provided reasonable data regarding the efficacy in lymphomas c) Early, retrospective data suggests that BEAM may be efficacious in MM however due to the lack of prospective controlled randomized clinical trial, there is adequate equipoise regarding its efficacy and moreover its comparative efficacy in relation to Melphalan and; D) there are known limitations in the standard-of-care for MM, Melphalan, namely, relatively low rates of complete response at the time of Autologous stem-cell transplantation (ASCT) and poor progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a new diagnosis of MM according to the International Myeloma Working Group (IMWG) working criteria undergoing autologous or syngeneic hematopoietic transplantation

   According to these criteria, the following must be met:
   1. Monoclonal plasma cells in the bone marrow > 10% (or proven plasmacytic infiltration in bone marrow biopsy) and/or presence of a biopsy-proven plasmacytoma.
   2. Monoclonal protein (M-protein) present in the serum and/or
   3. Myeloma-related organ dysfunction (1 or more) of the following. A variety of other types of end-organ dysfunctions can occasionally occur and lead to a need for therapy: - [C] Calcium elevation in the blood, defined as serum calcium > 10.5 mg/dl or upper limit of normal [R] Renal insufficiency (defined as serum creatinine above normal) [A] Anemia, defined as hemoglobin < normal - [B] Lytic bone lesions or osteoporosis. If a solitary (biopsy-proven) plasmacytoma or osteoporosis alone (without fractures) are the sole defining criteria, then > 30% plasma cells are required in the bone marrow
2. Patients must have received initial therapy for MM; at least 2 cycles with a minimum of partial response as defined by IMWG guidelines.
3. Age >=18, < 70years.
4. Karnofsky >70.
5. Life expectancy is not severely limited by concomitant illness based on the Hematopoietic Cell Transplant Comorbidity Index (HCT-CI) [8, 9] including:

   1. Left ventricular ejection fraction >50%. No uncontrolled arrhythmias or symptomatic cardiac disease.
   2. FEV1, FVC and DLCO >50%. No symptomatic pulmonary disease.
   3. HIV-negative.
   4. Bilirubin <2 mg/dl, SGPT <2.5 x normal.
   5. Creatinine clearance > 50 cc/min, estimated or measured.
6. Proficient in English
7. Signed informed consent

Exclusion Criteria:

1. Pregnant or lactating females
2. Limited verbal or reading English proficiency
3. Insufficient cognitive or comprehensive capability to provide informed consent
4. Uncontrolled infection
5. Planned tandem autologous/reduced intensity allograft
6. Insufficient peripheral blood stem cells (PBSC) in storage for an autologous transplant (<4.0 x 106 CD34+ cells/kg total).
7. Prior autologous transplant.
8. Patients unwilling to practice adequate forms of contraception if clinically indicated. Male patients on study need to be consulted to use latex condoms even if they have had a vasectomy every time they have sex with a woman who is able to have children
9. Patients with history of seizures
10. Prior history of another malignancy with a life expectancy of <3 years.
11. Known amyloidosis
12. Uncontrolled CNS myeloma
13. Anesthesia Society of America Physical Status (ASA PS) of 4 or greater

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 12 months
  Compare the complete response rates at the time of ASCT following either a high dose BEAM conditioning regimen or a monotherapy Melphalan conditioning regimen

SECONDARY OUTCOMES:
Hospitalization Duration | 12 months
  Measure and compare the duration of hospitalization exclusive of high dose regimen between arms
Progression Free Survival | 12 months
  Measure and compare the Progression Free Survival between study regimens
Overall Survival | 12 months
  Measure and compare the Overall Survival between study regimens

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States